CLINICAL TRIAL: NCT06696456
Title: An Evaluation of the Long Term Safety and Efficacy of AAVAnc80-hOTOF Gene Therapy in Individuals With Sensorineural Hearing Loss Due to Otoferlin Gene Mutations
Brief Title: Long Term Follow-up Study of AAVAnc80-hOTOF Gene Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Akouos, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: AK-OTOF-LTFU
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-01

CONDITIONS: Otoferlin Gene-mediated Hearing Loss
Keywords: Otoferlin; Deafness, autosomal recessive 9 (DFNB9); Hearing loss; Hearing loss, bilateral; Hearing loss, sensorineural; Auditory neuropathy (AN)
MeSH Terms: conditions — Deafness, Autosomal Recessive 9; Deafness; Hearing Loss; Hearing Loss, Bilateral; Hearing Loss, Sensorineural; Auditory neuropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Participants: Individuals with otoferlin gene-mediated hearing loss who received intracochlear administration of AAVAnc80-hOTOF in the AK-OTOF-101 Clinical Trial

SUMMARY:
This multi-center, observational, post-intervention long term follow-up (LTFU) study will monitor for safety and efficacy of AAVAnc80-hOTOF in individuals with sensorineural hearing loss due to otoferlin gene mutations who have previously received intracochlear administration of AAVAnc80-hOTOF in the AK-OTOF-101 Clinical Trial.

DETAILED DESCRIPTION:
After completing one year of initial safety and efficacy assessments following an intracochlear administration of AAVAnc80-hOTOF in AK-OTOF-101, participants will continue to be observed for an additional approximately four years of safety and efficacy follow-up in this LTFU study, for a total of approximately five years of safety and efficacy observations after vector administration. For each participant, evaluations in the LTFU study will occur at approximately one and a half years and two years after vector administration, followed by annual visits through Year 5; the duration in this LTFU study is approximately four years, with the aim of understanding and mitigating any risks related to delayed adverse events, as well as characterizing the durability of effect of the AAVAnc80-hOTOF.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with otoferlin gene-mediated hearing loss who received intracochlear administration of AAVAnc80-hOTOF in the AK-OTOF-101 Clinical Trial
* Legally authorized representative and/or participant willingness to comply with all study requirements, as evidenced by successful completion of the informed consent process or permission and participant assent process (where appropriate)

Exclusion Criteria:

* Any condition that would not allow the potential participant to complete follow-up examinations during the course of the study and/or, in the opinion of the Investigator, makes the potential participant unsuitable for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with otoferlin gene-mediated hearing loss who received intracochlear administration of AAVAnc80-hOTOF in the AK-OTOF-101 Clinical Trial.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2033-04 (Estimated); Study Completion 2033-04 (Estimated)

PRIMARY OUTCOMES:
Long term safety of AAVAnc80-hOTOF, including the incidence and frequency of late-occurring adverse events (AEs) | Through study completion, approximately four years.
  The following adverse events will be collected:
  1. The development of new or exacerbation of malignancies (oncologic), neurologic, rheumatologic or other autoimmune, hematologic disorders, or new infections (if the infection is potentially related to AAVAnc80-hOTOF
  2. AEs that are related to AAVAnc80-hOTOF and/or the administration procedure
  3. AEs of special interest
  4. All serious adverse events regardless of severity or of relationship to participation in the AK-OTOF-101 Clinical Trial

SECONDARY OUTCOMES:
Auditory Brainstem Response (ABR) Threshold | Through study completion, approximately four years.
  Changes in ABR intensity threshold (decibels normal hearing level [dB nHL])

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Reape, M.D., Study Director — Akouos, Inc.
Locations (4):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona, Spain
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AK-OTOF-101: Gene Therapy Trial for Otoferlin Gene-mediated Hearing Loss — https://clinicaltrials.gov/study/NCT05821959?cond=otoferlin&rank=3